CLINICAL TRIAL: NCT05986331
Title: A Randomized, Double-Blind Clinical Study of the Efficacy and Safety of BCD-201 (JSC BIOCAD) and Keytruda® in Patients With Unresectable or Metastatic Melanoma
Brief Title: Clinical Study of the Efficacy and Safety of BCD-201 and Keytruda in Subjects With Advanced Melanoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-201-2
Record Dates: First submitted 2023-02-13; First posted 2023-08-14 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-201 group (Experimental): BCD-201 200 mg as a 30-minute intravenous infusion once every 3 weeks
  Interventions: Drug: BCD-201
- Keytruda (Active Comparator): Keytruda 200 mg as a 30-minute intravenous infusion once every 3 weeks
  Interventions: Drug: Keytruda

INTERVENTIONS:
Drug: BCD-201 — up to 8 treatment cycles
  Other Names: Pembrolizumab
  Arms: BCD-201 group
Drug: Keytruda — up to 8 treatment cycles
  Other Names: pembrolizumab
  Arms: Keytruda

SUMMARY:
This clinical study is designed as a randomized, double-blind trial. Subjects with unresectable, metastatic, or recurrent skin melanoma will be randomized to one of the two study groups (BCD-201 group and Keytruda group) at a 1:1 ratio.

The goal of this study is to compare the efficacy and safety of BCD-201 and Keytruda as first-line therapy in subjects with unresectable, metastatic, or recurrent skin melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Histologically confirmed melanoma;
* Tumor first detected at the stage of advanced unresectable or metastatic disease, or disease progressing during or recurring after previous radical therapy;
* ECOG score 0-1;
* At least one measurable lesion according to RECIST 1.1;
* Laboratory test results consistent with adequate functioning of systems and organs;
* Willingness of men and women of childbearing potential to use highly effective contraceptive methods from the signing of the informed consent form, throughout the study and for 6 months after the administration of the last product dose.

Exclusion Criteria:

* Indications for radical therapy (surgery, radiation therapy);
* Uveal, ocular or mucosal melanoma;
* Active CNS metastases and/or carcinomatous meningitis;
* Subjects with severe concomitant disorders, life-threatening acute complications of the primary disease;
* Concomitant diseases and/or conditions that significantly increase the risk of AEs during the study;
* Active, known or suspected autoimmune disorders (subjects with type 1 diabetes mellitus or hypothyroidism requiring only hormone-replacement therapy and those with skin disorders [vitiligo, alopecia, or psoriasis] not requiring systemic therapy are eligible to participate);
* The need for therapy with glucocorticoids or any other drugs with immunosuppressive effects within 14 days prior to randomization;
* History of (non-infectious) pneumonitis requiring glucocorticoid therapy or pneumonitis at the time of screening;
* Hypersensitivity or allergy to any of the pembrolizumab product components;
* Pregnancy or breastfeeding, as well as intention to become pregnant or father a child during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare the overall response rate (ORR) in the BCD-201 group and the Keytruda group | 24 weeks of treatment
  ORR according to RECIST 1.1

SECONDARY OUTCOMES:
To compare the ORR according to iRECIST in the BCD-201 group and the Keytruda group | every 12 weeks up to 2 years
  ORR according to iRECIST
To compare the duration of response in the BCD-201 group and the Keytruda group | up to 2 years
  Duration of response will be calculated from the moment of registration of response till event (progression or death)
To compare the time to response according to RECIST 1.1 and iRECIST in the BCD-201 group and the Keytruda group | every 12 weeks up to 2 years
  time to response will be calculated from the randomization date
To compare the disease control rate in the BCD-201 group and the Keytruda group | up to 2 years
  The percentage of the participants who have a Complete Response, a Partial Response or a Stable DIsease
To compare the progression-free survival (PFS) per RECIST 1.1 and iRECIST in the BCD-201 group and the Keytruda group | up to 2 years
  The time from the date of randomization until progression of disease according to RECIST 1.1 / iRECIST criteria or death
To compare the overall survival in the BCD-201 group and the Keytruda group | up to 2 years
  The time from the date of randomization until death
To compare the incidence of Treatment-Emergent Adverse Events (Safety profiles of BCD-201 and Keytruda) | through study completion, an average of 2 years.
  Presence of any adverse events (AEs), presence of adverse reactions (ARs), presence of serious adverse reactions (SARs), presence of severe ARs (grade 3 or higher severity according to CTCAE v.5.0), presence of ARs leading to discontinuation of study therapy, presence of immune-mediated AEs
Area under the concentration-time curve (AUC(0-504)) | up to 24 weeks of the double-blind treatment period
  Area under the plasma concentration versus time curve in the time interval from 0 to 504 hours
AUC(0-∞) | up to 24 weeks of the double-blind treatment period
  Area under the plasma concentration versus time curve in the time interval from 0 to time infinity
Peak Plasma Concentration (Cmax) | up to 24 weeks of the double-blind treatment period
  maximum concentration of pembrolizumab
Time to maximum concentration (Tmax) | up to 24 weeks of the double-blind treatment period
  time to maximum concentration of pembrolizumab
Elimination rate constant (kel) | up to 24 weeks of the double-blind treatment period
  kel of pembrolizumab
Total clearance (Cl) | up to 24 weeks of the double-blind treatment period
  Cl of pembrolizumab
Steady-state volume of distribution of the drug substance (Vd) | up to 24 weeks of the double-blind treatment period
  Vd of pembrolizumab
Half-life period (T1/2) | up to 24 weeks of the double-blind treatment period
  T1/2 of pembrolizumab
Concentrations at the end of each infusion (CEOI) | up to 24 weeks of the double-blind treatment period
  concentrations at the end of each infusion of pembrolizumab
To compare the immunogenicity of BCD-201 and Keytruda. | pre-dose to day169 of the double-blind treatment period, 8 timepoints
  Development of binding and neutralizing antibodies to pembrolizumab

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Budgetary healthcare institution of the Omsk region "Clinical oncological dispensary", Omsk
  - "Saint Petersburg Clinical Research and Practice Center for Specialized Medical Care (Oncology)", Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "Saint Petersburg State University", Saint Petersburg

IPD SHARING:
Plan to Share IPD: No